CLINICAL TRIAL: NCT05593523
Title: Fluorescence-based Detection of Inflammation and Necrosis to Inform Surgical Decision-making and Enhance Outcomes
Status: Active, not recruiting | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2022-1070; 1R01GM145723-01 (NIH); Protocol Version 3/27/2025 (Other: UW Madison); A539714 (Other: UW Madison)
Record Dates: First submitted 2022-10-20; First posted 2022-10-25 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-04

CONDITIONS: Burn Wound
Keywords: imaging; detection; necrosis
MeSH Terms: conditions — Burns; Necrosis | interventions — Indocyanine Green

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — For Cohort 1, involving subjects with partial thickness burns, one 4 mm tissue biopsy (optional) will be collected from the center of the burn wound after SWIG imaging is performed. Optional blood draw for research purposes.
  For Cohort 2, up to two biopsies, one from the center of the burn wound and the other from a secondary location also within the tissue to be excised, will be taken at the time of surgery, or on the day of planned surgery in the event surgery was canceled due to unexpected healing (optional biopsy). Optional blood draw for research purposes.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Aim 1: Partial Thickness Burn Wounds: Participants with 1-30% total body surface area (TBSA) partial thickness burn wounds admitted to the University of Wisconsin (UW) Burn Center within 24 hours of burn injury and expected to be admitted for 3 days.
  Indocyanine green angiography (ICGA) fluorescence imaging immediately after administration of 7mg of ICG, and second window indocyanine green (SWIG) fluorescence imaging ~24 hours after administration of up to 5 mg/kg ICG of human burn wounds. ICGA within 72 hours of admission with the OnLume Clinical Imaging System (CIS). SWIG fluorescence imaging will also be performed perioperatively if applicable.
  Interventions: Drug: Indocyanine green (ICG); Device: Clinical Fluorescence Imaging Device
- Aim 2: Deep Partial or Full Thickness Burn Wounds: Participants with 1-30% total body surface area (TBSA) deep partial or full thickness burn wounds that will likely require surgery.
  ICGA fluorescence imaging immediately after administration of 7mg of ICG, and second window indocyanine green (SWIG) fluorescence imaging ~24 hours after administration of up to 5 mg/kg ICG of human burn wounds. Imaging will occur with the OnLume Clinical Imaging System (CIS).
  Interventions: Drug: Indocyanine green (ICG); Device: Clinical Fluorescence Imaging Device

INTERVENTIONS:
Drug: Indocyanine green (ICG) — ICG is a well, known, FDA-approved dye
Device: Clinical Fluorescence Imaging Device — OnLume Clinical Imaging System or Commercially-available FDA approved clinical fluorescence imaging device (SPY Elite fluorescence imaging system, SPY-PHI portable handheld imaging system, or EleVision IR platform (also known as VS3-IR system)
  Other Names: Asimov-MSK Imaging System; OnLume; SPY Elite; SPY-PHI; EleVision IR; VS3-IR

SUMMARY:
This study investigates fluorescence image-guided surgery to allow precise identification of necrotic tissue both preoperatively and intraoperatively in burn patients. Furthermore, it uses a multi-model approach to elucidate the localization of ICG in inflammation and necrosis to determine how this novel use of a well-known fluorescence marker can be optimized to aid in surgical decision making. This proposal will provide the necessary data to support the design of a larger clinical trial to study the feasibility and efficacy of this technology to improve the precision of necrosis detection and removal and improve wound healing outcomes. Up to 100 participants will be on study for up to approximately 24 days.

DETAILED DESCRIPTION:
Tissue necrosis is a form of cell death caused by a wide variety of diseases and injuries. Current methods of detecting tissue necrosis to guide surgical decision making are limited. In burn injury, clinical visualization of tissue necrosis is the standard of care; however, it is an imprecise method that can result in delays in care, unnecessary surgery, and removal of viable tissue. There is a critical need to identify novel methods to improve the detection of necrosis in burn injury to aid perioperative clinical decision making. While Indocyanine Green Angiography (ICGA) has been shown to identify burn depth using perfusion as a surrogate marker for necrosis, it has not been widely adopted for clinical decision making. Recently, clinical trials using delayed imaging of high dose ICG (Second Window Indocyanine Green - SWIG) have shown promise in image-guided surgical resection of tumors. The investigators propose that SWIG imaging can be employed to enhance surgical decision-making in burn injury, as well as in many disease processes involving necrosis. The knowledge gained from this project will fill the critical need to prevent unnecessary surgery, improve surgical precision, and provide insight into ICG localization in inflamed and necrotic tissue.

The goal of this project is to characterize the SWIG fluorescence in burn inflammation and necrosis on a macroscopic and microscopic level.

Cohort 1 - The investigators will characterize fluorescent signals from SWIG in the healing potential of indeterminate depth burns in humans.

Cohort 2 - The investigators will examine the association between SWIG fluorescence and depth of necrosis in surgically excised burns, and in cases where surgery is canceled due to unexpected healing, in human subjects.

This project will result in clinical data testing of ICG for direct detection of necrotic tissue using a fluorescence imaging device optimized for burn surgery, while developing a platform for quantification of tissue necrosis and characterization of ICG-avid necrosis. These studies will provide necessary data to inform the design of a larger clinical trial to determine the efficacy and validity of ICG fluorescence-guided clinical decision making to improve outcomes for burn patients.

ELIGIBILITY:
Inclusion Criteria:

* English speaker
* Patients with partial thickness indeterminate depth burn wounds that occurred within 24 hours of admission and are expected to require admission for at least 3 days (Aim 1) or with deep partial thickness or full thickness burn wounds that are 1-30% TBSA and will likely require surgery (Aim 2)
* Subject understands the study procedures and can provide informed consent to participate in the study and authorization for release of relevant protected health information to the study investigator

Exclusion Criteria:

* Contraindication to Indocyanine Green (ICG) injection, i.e. previous reaction to ICG (adverse event rate: 1 in 42,000) or Iodine allergy.
* Inability to obtain consent
* Subject with pre-existing inflammatory diseases or chronically treated before admission to the hospital with steroids or nonsteroidal anti-inflammatory drugs or biologics
* Subject with immune deficiency (HIV infection or use of corticosteroids, cytostatic drugs, tetracycline and certain bisphosphonates)
* Subject with known or suspected infections or on antibiotic therapy
* Subject known or suspected to be pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Aim 1: Human subjects with partial thickness burn wounds admitted to the UW Burn Center within 24 hours of burn injury and expected to be admitted for 3 days Aim 2: Human subjects with 1-30% total body surface area (TBSA) deep partial or full thickness burn wounds that require surgery.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-03-09 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Signal to Background Ratio (SBR) of ICGA and SWIG Fluorescence Images | up to 96 hours after injury (up to 4 days on study)
  Quantitative assessment of all ICGA and SWIG fluorescence images will be achieved in part by measuring the fluorescence signal-to-background ratio (SBR).
Standard Deviation of ICGA and SWIG Fluorescence Images | up to 96 hours after injury (up to 4 days on study)
  Quantitative assessment of all ICGA and SWIG fluorescence images will be achieved in part by measuring the fluorescence standard deviation.
Spatial Pattern of ICGA and SWIG Fluorescence Images | up to 96 hours after injury (up to 4 days on study)
  Qualitative characterization of all ICGA and SWIG fluorescence images will be achieved by evaluating the fluorescence spatial patterns and features.
Burn Surgeon Assessment of Wound Healing (Yes/No) | up to 24 days from burn injury (up to 21 days on study)
  For Aim 1, a burn surgeon blinded to the fluorescence data will perform an assessment of complete wound healing without surgery (Yes/No) at 21 ± 3 days from burn injury.
Burn Surgeon Assessment of Graft Loss (Yes/No) | up to 21 days after discharge following skin grafting (up to 31 days on study)
  For Aim 2, a burn surgeon blinded to the fluorescence data will perform an assessment of presence or absence of graft loss (Yes/No) 14 ± 7 days after discharge following skin grafting.
Depth of Necrotic Tissue as a Percentage of the Tissue Biopsy Thickness | sample collected up to 4 days on study

SECONDARY OUTCOMES:
Spatial Correlation of ICG fluorescence and Cell Necrosis and Inflammation | sample collected up to 4 days on study

CONTACTS AND LOCATIONS:
Overall Officials: Angela Gibson, MD, PHD, Principal Investigator — University of Wisconsin - Madison School of Medicine and Public Health
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No